CLINICAL TRIAL: NCT04529694
Title: Patient Characteristics and Cognitive Behavior Therapy for Depression
Brief Title: Patient Characteristics and Cognitive vs. Behavioral Therapies for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Daniel R. Strunk, Associate Professor of Psychology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011B0342
Record Dates: First submitted 2020-08-14; First posted 2020-08-28 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-only Intervention (Active Comparator): This condition includes cognitive interventions drawn from cognitive therapy as described in Beck, Rush, Shaw, & Emery (1979).
  Interventions: Other: Psychotherapy
- Behavioral-only Intervention (Active Comparator): The condition includes behavioral interventions drawn from cognitive therapy as described in Beck, Rush, Shaw, & Emery (1979).
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy

SUMMARY:
This is a retrospective registration. The study was conducted at The Ohio State University from 2011 to 2012. This study was approved by an Institutional Review Board at The Ohio State University. The investigators retroactively registered this trial to facilitate publishing results in journal that now require registration. Any reference to the study's registration will make it clear that the registration was retroactive. Cognitive behavior therapy (CBT) has been shown to be an effective treatment for depression. However, a substantial number of patients do not respond to treatment or continue to be symptomatic at its conclusion. An important goal of ongoing research is to find ways to enhance treatment outcomes. One approach to doing this is to modifying existing treatments to individualize the approach to better meet the needs of individual patients. In this study, the investigators tested two main components of CBT to empirically evaluate patient characteristics that may predict differential response to these components. By using components of CBT, any suggestions about the strategies that are best suited to different patients are likely be easily implemented by therapists providing CBT. The two treatment components the investigators examined were: cognitive interventions (e.g., challenging negative automatic thoughts) and behavioral interventions (e.g., engaging in activities to promote a sense of pleasure or accomplishment). The investigators recruited adults with major depressive disorder and randomized them to a cognitive or behavioral intervention. After 8 weeks of treatment, patients were randomized again to a cognitive or behavioral intervention. Consequently, participants were offered a total of 16 weeks of treatment. Depressive symptoms were assessed with the Beck Depression Inventory-II (BDI-II) and the Hamilton Rating Scale for Depression (HRSD), with the latter being the primary outcome measure. Several variables that might serve to predict differential response to cognitive and behavioral treatments were also assessed. The results of this study may help to elucidate how cognitive or behavioral interventions might be selected so as to enhance overall treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder (MDD) according to DSM-IV criteria (APA, 1994)
* Able and willing to give informed consent

Exclusion Criteria:

* History of bipolar affective disorder or psychosis
* Current Axis I disorder other than MDD if it constitutes the predominant aspect of the clinical presentation and if it requires treatment other than that being offered
* History of substance dependence in the past six months
* Subnormal intellectual potential (IQ below 80, testing to be initiated if clinically indicated)
* Clear indication of secondary gain (e.g., court ordered treatment)
* Current suicide risk or significant intentional self-harm in the last six months sufficient to preclude treatment on an outpatient basis
* If clients currently being treated with a medication for depression: (1) no change in medication and a stable dose for at least 1 month prior to their initial assessment; and (2) agreeing to not make changes to medication or medication dose during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10-20 (Actual); Primary Completion 2012-06-26 (Actual); Study Completion 2012-06-26 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale for Depression at week 8 and week 16 | Time Frame: Weeks 0-8 and 0-16, assessments occurred at weeks 0, 4, 8, and 16.
  The Hamilton Rating Scale for Depression is a 17-item interviewer evaluated assessment of depressive symptoms. Scores range from 0 to 52, with higher scores indicating greater depressive symptoms.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory-II at week 8 and week 16 | Time Frame: Weeks 0-8 and 0-16, assessments occurred at every session through week 16.
  The Beck Depression Inventory-II is a 21-item self-report measure of depressive symptoms. Scores range from 0 to 63, with higher scores indicating greater depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We will consider requests for data sharing, pending approval from our IRB.

REFERENCES:
- [Derived] Murphy ST, Cooper AA, Hollars SN, Strunk DR. Who Benefits From a Cognitive vs. Behavioral Approach to Treating Depression? A Pilot Study of Prescriptive Predictors. Behav Ther. 2021 Nov;52(6):1433-1448. doi: 10.1016/j.beth.2021.03.012. Epub 2021 Apr 9. PMID 34656197